CLINICAL TRIAL: NCT01251315
Title: PILOT: The Effects of Short Term Administration of a Novel Glutathione Precursor (FT061452), on Serum and Intracellular Glutathione Levels
Brief Title: The Effects of a Glutathione Precursor (FT061452),on Serum and Intracellular Glutathione Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Naureen Tareen, Principal Investigator, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10 - 04 - 2268 - 01
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Oxidative Stress
Keywords: Glutathione; Antioxidant; Free radical; Oxidative stress; N-Acetyl Cysteine; Glutathione precursor
MeSH Terms: interventions — Cellulose; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo low dose (Placebo Comparator): Placebo for low dose group given as a single dose.
  Interventions: Drug: Placebo low dose
- N Acetyl cysteine, 600mg (low dose) (Active Comparator): N-Acetyl Cysteine (NAC)600 mg (low dose) given as a single dose.
  Interventions: Drug: N Acetyl cysteine, 600mg (low dose)
- Proimmune 200(FT061452) (Active Comparator): Proimmune 200(FT061452) low dose group 3000 mg given as a single dose.
  Interventions: Drug: Proimmune 200 (FT061452) 3000mg low dose
- Placebo high dose (Placebo Comparator): Placebo given to high dose group given as a single dose.
  Interventions: Drug: Placebo (high dose)
- N Acetyly cysteine, 1200mg (high dose) (Active Comparator): N-Acetyl Cysteine(NAC)1200mg (high dose) given as a single dose.
  Interventions: Drug: N Acetyl cysteine, 1200mg (high dose)
- FT061452, 6000mg high dose (Active Comparator): Proimmune 200(FT061452) high dose group given 6000 mg as a single dose.
  Interventions: Drug: FT061452, 6000mg high dose

INTERVENTIONS:
Drug: Placebo low dose — This is a prospective randomized controlled pilot study, which will include twenty-four (24) healthy individuals.The first 12 subjects (low dose) will be randomized into three sub groups. The first group will be given a single dose of placebo.
  Other Names: Cellulose
  Arms: Placebo low dose
Drug: N Acetyl cysteine, 600mg (low dose) — The sub-group of four subjects (low dose) will be given a single dose of 600 mg of N-Acetyl Cysteine (NAC).
  Other Names: NAC
  Arms: N Acetyl cysteine, 600mg (low dose)
Drug: Proimmune 200 (FT061452) 3000mg low dose — The sub-group of four subjects (low dose) will be given a single dose of Proimmune 200 (FT061452) 3000mg low dose'
  Other Names: Proimmune-200 (FT061452)
  Arms: Proimmune 200(FT061452)
Drug: Placebo (high dose) — The second sub set of 12 subjects (high dose) will be randomized into three sub groups. The first group will be given a single dose of placebo.
  Other Names: Cellulose
  Arms: Placebo high dose
Drug: N Acetyl cysteine, 1200mg (high dose) — N Acetyl cysteine (high dose) N-Acetyl Cysteine(NAC)1200mg (high dose) given as a single dose.
  Other Names: NAC
  Arms: N Acetyly cysteine, 1200mg (high dose)
Drug: FT061452, 6000mg high dose — Proimmune 200(FT061452) high dose group given 6000 mg as a single dose.
  Other Names: Proimmune-200 (Glutathione precursor)
  Arms: FT061452, 6000mg high dose

SUMMARY:
Glutathione is a powerful protective substance found within every cell in the body. It has been shown that glutathione levels go down as a person gets older, which makes a person more likely to get heart disease, high blood sugar problems and different kind of cancers. N-Acetyl Cysteine is used as a dietary supplement. It has been reported to increase glutathione levels in the body. The diet supplement called ProImmune is also changed by the body into glutathione. Therefore, the purpose of this study is to find out the effect of ProImmune in healthy people. This study will also help to prove whether or not the ProImmune is able to improve the blood levels of glutathione in healthy people.

DETAILED DESCRIPTION:
Glutathione (gamma-glutamyl-cysteine-glycine; GSH) is a powerful antioxidant found within every cell. GSH is predominantly known to protect the cells from damage caused by free radicals. The concentration of glutathione declines with age, stress, and in some age-related diseases. When glutathione becomes deficient, a series of events are initiated termed "oxidative stress" and the associated cell signaling leads to impaired immune function and similar abnormalities in numerous cell systems.

Oral glutathione is ineffective in replenishing glutathione levels and reversing the abnormal signaling pathways associated with oxidative stress. Intravenous glutathione has been shown to be effective but is short-lived. N-Acetyl Cysteine, a glutathione precursor, has had limited efficacy in clinical settings and suffers from an adverse effect profile.Null Hypothesis (primary): The administration of FT061452 will not increase serum and intracellular glutathione levels in comparison to N-Acetyl Cysteine (NAC), and placebo.

Null Hypothesis (secondary): The administration of FT061452 will not improve vascular function in comparison to N-Acetyl Cysteine (NAC), and placebo.

The Specific Aims of this pilot study are to:

* Compare the change in serum and intracellular glutathione levels following the administration of a novel oral glutathione precursor, FT061452, (modified glutathione with selenium added, and cystine replacing cysteine, in doses equivalent to NAC) compared to low dose or usual dose of NAC, and placebo.
* Compare the change in select clinical parameters (vascular function) following the administration of a novel oral glutathione precursor, FT061452, (modified glutathione with selenium added, and cystine replacing cysteine) compared to N-Acetyl Cysteine (NAC), and placebo.
* As a pilot study a third goal is to generate effect sizes for appropriately powering future clinical trials.

Background:

Increased rates of adverse health outcomes for racial and ethnic minorities have been linked to a confluence of socio-cultural, environmental, immunological, and genetic based factors, frequently acting in concert. Ultimately, the majority of these factors lead to adverse physiologic and cellular changes. However, it is the chronic activation of these neurohormonal systems through the above stresses that lead to maladaptive health consequences such as accelerated apoptosis, atherogenesis, altered immune function, and other dysregulations of cellular function. Ultimately, stress related cellular activities contribute to many of the observed premature chronic diseases in humans, many of which are found in disproportionately high rates in minority communities. Glutathione is the major regulator of the cellular oxidative state that buffers many of these stress related pathways. When glutathione becomes deficient there occurs an increase in reactive oxidative species (ROS) that collectively can be termed "oxidative stress". Clinically, oral glutathione (GSH) has been ineffective in replenishing glutathione levels and reversing the associated abnormal cellular signaling. GSH as a whole molecule cannot be taken up by cells in mammals but is largely metabolized in the gastrointestinal tract into constituent amino acids, including the highly oxidizable L-cysteine, which cannot be re-united extracellularly into glutathione as its re-assimilation requires two cytosolic, ATP-dependent enzymes. Thus, the processes that achieve glutathione synthesis require special conditions that are only present within the cell. Oral glutathione preparations are limited by their ability to provide adequate substrate to stimulate intracellular glutathione synthesis due to L-cysteine being highly oxidizable. Intravenous glutathione administration is expensive, short-lived, and impractical, as the transiently higher plasma concentrations are largely independent of intracellular glutathione activity, where much of the oxidative balance is performed. N-Acetyl Cysteine (NAC), a glutathione precursor, has had limited efficacy in clinical settings and suffers from an adverse side-effect profile. However, preliminary findings of a novel glutathione precursor with vitamin implications (FT061452) indicate it can affect the metabolism of glutathione via 2 mechanisms: 1) increasing the availability of intracellular cysteine by using the more stable cystine as the physiologic and more stable cysteine carrier which can traverse the cell membrane and create a more optimal Cys/CySS redox state, and 2) adding selenium, an important co-factor for glutathione reductase. Thus, FT061452 appears to provide a greater cellular delivery of substrate to attenuate oxidative stress, in comparison to traditional glutathione precursors, which despite showing promise,have not demonstrated consistent clinical efficacy.

Preliminary studies ; Preliminary studies to investigate GSH and several GSH analogs might protect spermine-induced apoptosis in aortic vascular smooth muscle cells (VSMC) have been promising. Given that spermine (a uremic toxin) increases intracellular ROS and promotes apoptosis in some cultured cells, we first examined the generation of ROS along with intracellular levels of reduced GSH and the ratio of reduced GSH and oxidized glutathione (GSH/GSSG) in VSMC in response to spermine treatment and its attenuation by concomitant administration of similar strengths of GSH, NAC and FT061452. While concomitant exposure of these cells to NAC, GSH, or FT061452 attenuated spermine-induced decrease in GSH levels, only the addition of the novel glutathione precursor, FT061452, to spermine treated cells increased intracellular GSH levels above control values.

Study Design & Method:

This is a prospective randomized controlled pilot study, which will include twenty-four (24) healthy individuals between ages of 30-65 years old. The study will occur over the course of two days. On Day 1, potential subjects will be screened to determine eligibility by mini history and physical exam, complete blood count (CBC) and complete metabolic panel (CMP). On Day 2, eligible subjects will report to Participant and Clinical Interactions Resource Center (formerly known as the CRC) after fasting overnight. The first 12 subjects (low dose) will be randomized into three groups, 1) those given a single dose of placebo, 2) those given 600 mg (low dose) of N-Acetyl Cysteine (NAC) or 3) those given 3000 mg of study drug (FT061452). Serum and intracellular glutathione levels, biomarkers, and non-invasive measures of vascular function were assessed at baseline, 2, 4 and 6 hours. During their stay in CRC, subjects in every group will be fed the same meal. The second 12 subjects (usual dose) will be randomized into three groups, 1) those given a single dose of placebo, 2) those given 1200 mg (usual dose) of N-Acetyl Cysteine (NAC) or 3) those given 6000 mg of study drug (FT061452). Serum and intracellular glutathione levels, biomarkers, and non-invasive measures of vascular function will be assessed at baseline, 2, 4 and 6 hours. During their stay in CRC, subjects in every group will be fed the same meal.

At baseline, 2, 4 and 6 hours, a blood sample (15 cc per draw) will be obtained for serum and intracellular glutathione levels, stored serum for biomarkers, and non-invasive measures of vascular function will be assessed at baseline and 6 hours, as follows: 1) Pulse wave velocity and Augmentation Index (via SphygmoCor): (central artery pressure and central aortic pulse pressure) and 2) Peripheral vascular endothelial function (via EndoPat): (% flow mediated dilation).

This study has potential benefits to others. The knowledge gained will provide realistic and practical information that guides the implementation of a non-pharmacological intervention to reduce the progression of age related morbidities. Because CDU's community is largely minority, the community of color will be included in this recruitment. The IRB exercises oversight of all protocols involving human subjects, monitors for adverse events, and performs audits of all approved protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be healthy male or female, 30 to 65 years of age.
2. Subjects must have a BMI between 20 and 35.
3. Subjects must be able to provide informed consent after risks and benefits have been explained.
4. Subjects must be non-smoking (defined as a subject who has not smoked for ≥ 6 months), and must agree to abstain from caffeine 72 hours prior to study day.
5. Subjects are in generally good health, based on pre-study medical history, physical examination and routine laboratory tests.
6. Subjects have, in the Investigator's opinion, no clinically significant disease and/or clinically significant abnormal laboratory values as determined by the Investigator based on medical history, physical examination, or laboratory evaluations conducted at the screening visit or on admission to the clinic.

Exclusion Criteria:

1. Subjects who have a history of drug or alcohol abuse within 6 months of study screening, as determined by the Investigator.
2. Subjects who have participated in any investigational trial within 30 days or six half-lives of the test drug's biologic activity, whichever is longer, before the start of the study (time of first dose).
3. Subjects who have clinically significant medical or psychiatric illnesses currently or within 30 days of start of study (time of first dose), as determined by 3. the Investigator.
4. Subjects who have had symptoms of any significant acute illness within 30 days prior to the start of study (time of first dose),
5. Subjects who have any condition that interferes with their ability to understand or comply with the requirements of the study.
6. Females who are pregnant or nursing or have a high likelihood of becoming pregnant during the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naureen Tareen, MD, Principal Investigator — Charles Drew University
Locations (1):
- Charles Drew University, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited between may 2010 through June 2010. Healthy volunteers were recruited by physician referrals from community clinics.
Pre-assignment Details: No enrolled participants were excluded.
Groups:
- Placebo Low Dose Group, Given Oral as a Single Dose: Placebo low dose group, given oral as a single dose
- N Acetyl Cysteine (Low Dose, 600mg Oral as a Single Dose): N Acetyl cysteine (low dose, 600mg oral as a single dose)
- Proimmune 200 (Low Dose, 3000 mg Oral as a Single Dose): Proimmune 200 (low dose, 3000 mg oral as a single dose)
- Placebo High Dose Group, Given Oral as a Single Dose: Placebo high dose group, given oral as a single dose
- N Acetyl Cysteine (High Dose, 1200 mg Oral as a Single Dose): N Acetyl cysteine (high dose 1200 mg oral as a single dose)
- Proimmune 200 (High Dose, 6000 mg Oral as a Single Dose): Proimmune 200 (high dose, 6000 mg oral as a single dose)
Period: Overall Study
Arm/Group | Placebo Low Dose Group, Given Oral as a Single Dose | N Acetyl Cysteine (Low Dose, 600mg Oral as a Single Dose) | Proimmune 200 (Low Dose, 3000 mg Oral as a Single Dose) | Placebo High Dose Group, Given Oral as a Single Dose | N Acetyl Cysteine (High Dose, 1200 mg Oral as a Single Dose) | Proimmune 200 (High Dose, 6000 mg Oral as a Single Dose)
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo-A: low dose oral x1
- N Acetyl Cysteine-A: N Acetyl cysteine low dose group (600mg oral X1)
- Proimmune 200-A: Proimmune 200 low dose group (3000mg oral X 1)
- Placebo-B: High dose oral X1
- N Acetyl Cysteine-B: N Acetyl Cysteine High dose group ( 1200mg oral X1)
- Proimmune 200-B: Proimmune 200 High dose group (6000mg oral x1)
- Total: Total of all reporting groups
Arm/Group | Placebo-A | N Acetyl Cysteine-A | Proimmune 200-A | Placebo-B | N Acetyl Cysteine-B | Proimmune 200-B | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (6.4) | 38.2 (3.8) | 45.5 (12.9) | 39.3 (6.8) | 38.0 (5.8) | 42.5 (9.2) | 40 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 3 | 1 | 2 | 10
  Male | 3 | 3 | 2 | 1 | 3 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 24

OUTCOME MEASURES:

1. Secondary Outcome: Augmentation Index
Description: Augmentation index (%) is defined as the percentage of the central pulse pressure which is attributed to the reflected pulse wave and, therefore, reflects the degree to which central arterial pressure is augmented by wave reflection" if appropriate augmentation index has been shown to be a predictor of adverse cardiovascular events in a high risk patient populations,higher augmentation index is associated with target organ damage. Absolute change of augmentation index from baseline to 6 hours will be estimated for the analysis.
Time Frame: Baseline and 6 hours
Measure: Mean (Standard Deviation); unit: percentage of the central pulse pressure
Groups:
- Placebo-A: Placebo low dose group
- N Acetyl Cysteine-A: N Acetyl cysteine low dose group ( 600mg oral x1)
- Proimmune 200-A: Proimmune 200 low dose group ( 3000mg oral x1)
- Placebo-B: Placebo High dose group
- N Acetyl Cysteine-B: N Acetyl Cysteine High dose group (1200 mg oral x1)
Arm/Group | Placebo-A | N Acetyl Cysteine-A | Proimmune 200-A | Placebo-B | N Acetyl Cysteine-B | Proimmune 200-B
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
percentage of the central pulse pressure
  Baseline | 20 (5.0) | 19.8 (10.2) | 28.5 (12.7) | 27 (10.8) | 20.3 (11.9) | 26.5 (6.0)
  6 hour | 11.3 (8.4) | 11.3 (6.9) | 19 (10.4) | 24.8 (5.3) | 17.5 (15.7) | 19.3 (6.6)

2. Primary Outcome: Intracellular Glutathione Level
Description: Mean intracellular glutathione level every 2 hour
Time Frame: 6 hours
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- N Acetyl Cysteine-A: N Acetyl cysteine low dose group
- Proimmune 200-A: Proimmune 200 low dose group
- N Acetyl Cysteine-B: N Acetyl Cysteine High dose group
- Proimmune 200-B: Proimmune 200 High dose group
Arm/Group | Placebo-A | N Acetyl Cysteine-A | Proimmune 200-A | Placebo-B | N Acetyl Cysteine-B | Proimmune 200-B
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
µmol/L
  Baseline | 221.5 (133.7) | 118.5 (131.2) | 508.5 (493.3) | 358.0 (116.9) | 147.8 (86.8) | 132.8 (168.3)
  2 hour | 242.3 (163.7) | 121.8 (120.4) | 342.8 (283.6) | 347.8 (109.5) | 149.5 (74.0) | 311.8 (228.7)
  4 hour | 178.0 (146.8) | 149.8 (167.1) | 440.8 (419.9) | 383.8 (159.2) | 133.5 (75.4) | 279.8 (228.7)
  6 hour | 236.5 (221.3) | 103.5 (104.0) | 317.8 (553.3) | 355.0 (319.4) | 125.0 (50.2) | 274.0 (240.6)

ADVERSE EVENTS:
Groups:
- Placebo-A: low dose group
- Placebo-B: High dose group
Arm/Group | Placebo-A | N Acetyl Cysteine-A | Proimmune 200-A | Placebo-B | N Acetyl Cysteine-B | Proimmune 200-B
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No